CLINICAL TRIAL: NCT05461716
Title: Incidence of Hypoglycemia Events in Patients With Stable Insulin-treated Type 2 Diabetes Mellitus: Continuous Glucose Monitoring vs. Self-Monitored Blood Glucose
Brief Title: Incidence of Hypoglycaemia Events in Patients With Stable Insulin-treated Type 2 Diabetes Mellitus Based on Continuous Glucose Monitoring
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: George E. Dafoulas (Other)
Collaborators: Centre for Research and Technology Hellas (Other); University of Ioannina (Other)
Responsible Party: Sponsor-Investigator, George E. Dafoulas, Clinical Research Fellow, University of Thessaly
Organization: University of Thessaly (Other)
Other Study IDs: 857223-UC3GR
Record Dates: First submitted 2022-07-12; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus Type 2 With Hypoglycemia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: periodic use of Continuous Glucose Monitoring (CGM) — Identification of hypoglycaemia events, based on use of Continuous Glucose Monitoring (CGM) for at least 14days, in subgroups of T2DM patients with high risk of hypoglycaemia

SUMMARY:
Certain groups of patients with Type 2 Diabetes Mellitus (T2DM) appear to have higher risk of hypoglycaemia. Periodic use of Continuous Glucose Monitoring (CGM), has been suggested as a method to detect hypoglycaemia events in certain subgroups of patients with high risk of hypoglycaemia.

The aim of the present study is to contribute to the identification of subgroups of T2DM patients with high risk of hypoglycemia events, based on periodic use of Continuous Glucose Monitoring (CGM).

DETAILED DESCRIPTION:
Some studies successfully achieved standard glycemic targets without increased hypoglycaemia in older adults and other groups of patients with high risk of hypoglycaemia events.

However these trials usually exclude adults with poor health and comorbidities, when they support the concept that intensive strategies for selected individuals can be effective and safe. The compendium of results from these and other published analyses suggests that although some patients may benefit from tighter targets, many are unable to reach these targets, and aggressive therapy may be harmful to some patients without the benefit of reducing complications.

Although avoidance of hypoglycaemia is a critical treatment strategy, overall glucose control remains an important goal. The present treatment guidelines fail to locate the proper subgroup of patients with Type 2 Diabetes Mellitus (T2DM), that could be benefited of glycemic control balanced with the adverse effects of glucose-lowering medications and a patient's age, overall health status, and functional and intellectual capacity. The aim of the present study is to contribute to the identification of subgroups of T2DM patients with high risk of hypoglycemia events, based on periodic use of Continuous Glucose Monitoring (CGM).

ELIGIBILITY:
Inclusion Criteria:

* being older than 40 years of age
* having type 2 diabetes for at least 1 year
* being on insulin therapy for at least 3 months before recruitment
* having the ability to perform self-monitoring
* being able to wear a CGM system during 2 weeks
* having a stable metabolic situation, defined as having no need to add new treatments or make any changes in insulin dosage of more than 10% in the preceding 2 months

Exclusion Criteria:

* Having severe hearing or vision problems or any other acute or chronic condition that would limit the ability of the user to participate in the study
* Being institutionalised or person not capable of giving consent
* Pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Primary Care Services or the Outpatient Department of the Hospital
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Detection of hypoglycaemic events | frequency of hypoglycemia using the 12-week self-monitored blood glucose (SMBG) measurement profile and the 2 CGM weeks

SECONDARY OUTCOMES:
Glucose Management Indicator (GMI) correlation with HbA1c | 12 weeks self-monitored blood glucose (SMBG) measurement profile and the 2 CGM weeks
Glycaemic control (Time in Range) | 12 weeks self-monitored blood glucose (SMBG) measurement profile and the 2 CGM weeks
EQ5D (Generic HRQL) | 12 weeks self-monitored blood glucose (SMBG) measurement profile and the 2 CGM weeks
  Generic Health Related Quality of Life (HRQL)
Problem Areas in Diabetes scale - PAID (Disease specific HRQL) | 12 weeks self-monitored blood glucose (SMBG) measurement profile and the 2 CGM weeks
Assess the risk of hypoglycemia with Hypoglycemia Patient Questionnaire | 12 weeks self-monitored blood glucose (SMBG) measurement profile and the 2 CGM weeks
Registry of hypoglycaemia events in patients with T2DM treated with insulin and insulin secretagogues | 12 weeks self-monitored blood glucose (SMBG) measurement profile and the 2 CGM weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology and Metabolic Diseases, University Hospital of Larisa, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No
The IPD are going to be shared within the provisions of the European Commission Grant Agreement and Consortium Agreement of the Study

REFERENCES:
- [Background] Pazos-Couselo M, Garcia-Lopez JM, Gonzalez-Rodriguez M, Gude F, Mayan-Santos JM, Rodriguez-Segade S, Rodriguez-Garcia J, Casanueva F. High incidence of hypoglycemia in stable insulin-treated type 2 diabetes mellitus: continuous glucose monitoring vs. self-monitored blood glucose. Observational prospective study. Can J Diabetes. 2015 Oct;39(5):428-33. doi: 10.1016/j.jcjd.2015.05.007. Epub 2015 Aug 5. PMID 26254702
- [Background] Seaquist ER, Anderson J, Childs B, Cryer P, Dagogo-Jack S, Fish L, Heller SR, Rodriguez H, Rosenzweig J, Vigersky R. Hypoglycemia and diabetes: a report of a workgroup of the American Diabetes Association and the Endocrine Society. Diabetes Care. 2013 May;36(5):1384-95. doi: 10.2337/dc12-2480. Epub 2013 Apr 15. PMID 23589542